CLINICAL TRIAL: NCT00671320
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group Study To Compare The Efficacy And Tolerability Of Valdecoxib Vs. Diclofenac In Ankle Sprain
Brief Title: A Multi-Center, Randomized, Double-Blind, Parallel Group Study To Compare The Efficacy And Tolerability Of Valdecoxib And Diclofenac In Patients With A Sprained Ankle
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VALA-0513-146; A3471037
Record Dates: First submitted 2008-03-31; First posted 2008-05-05 (Estimated); Last update posted 2008-05-05 (Estimated); Status verified 2008-04

CONDITIONS: Pain; Sprains and Strains; Sprain
Keywords: acute ankle sprain, acute pain, South America
MeSH Terms: conditions — Pain; Sprains and Strains; Acute Pain | interventions — valdecoxib; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib
- Arm 2 (Active Comparator)
  Interventions: Drug: diclofenac

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 40 mg tablet by mouth twice daily (BID) on Day 1 and then once daily (QD) on Days 2 to 7
  Arms: Arm 1
Drug: diclofenac — diclofenac 75 mg capsule by mouth twice daily (BID) for 7 days
  Arms: Arm 2

SUMMARY:
To determine whether valdecoxib 40 mg twice a day the first day and then 40mg once a day until Day 7, was at least as effective as diclofenac 75 mg twice a day for 7 days, in treating acute first or second degree ankle sprain. The study also compared valdecoxib and diclofenac with respect to time to onset of pain relief (measured after the first dose), tolerability (adverse events) and time to return to Normal Function/Activity, among other measures.

ELIGIBILITY:
Inclusion Criteria:

* Patients had sprained their ankle within 48 hours
* The sprain was a first or second degree ankle sprain of the lateral aspect, specifically: anterior talofibular ligament and/or calcaneofibular ligament
* At presentation patients were to have had moderate-severe ankle pain, (i.e., patient's assessment of ankle pain, on full weight bearing, using a 100 mm visual analog scale (VAS) was ≥ 45 mm), have a minimum rating of 2 on the Patient's Global Assessment of Ankle Injury and Patient's Assessment of Normal Function/Activity
* Investigator must have thought that the patient required and was eligible for therapy with an anti-inflammatory agent and/or analgesic to control symptoms

Exclusion Criteria:

* Women who were not post-menopausal or surgically sterilized, or who had have a positive urine pregnancy test prior to randomization and/or were not using adequate contraception according to the judgment of the Investigator
* Patients with a similar injury of the same joint within the last 6 months
* Clinical evidence of complete rupture of ankle ligaments (third degree sprain), required bed rest, hospitalization, surgical intervention for the ankle injury or non-removable full cast, bilateral occurrence of ankle injury or ankle and knee injury on the same side
* Patients with esophageal, gastric or duodenal ulcer within 30 days prior to randomization or had active GI or other disease that in the opinion of the investigator would preclude safe participation by the subject in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2002-12; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Patient's assessment of ankle pain VAS | Day 4

SECONDARY OUTCOMES:
Time to onset of pain relief | 0, 15, 30, 45, and 60 minutes after first dose
Physician's global assessment of ankle injury | Days 1, 4, and 7
Patient's global assessment of ankle injury | Days 1, 4 and 7
Patient's assessment of normal function/activity | Days 1 to 7
Patient's and physician's satisfaction assessments | Day 7
Patient's assessment of ankle pain on visual analogue scale (VAS) | Days 1 to 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Argentina (3):
  - Pfizer Investigational Site, Avellaneda, Buenos Aires
  - Pfizer Investigational Site, San Isidro, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
- Chile (2):
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Santiago
- Colombia (6):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Bogotá, Cundinarmarca
  - Pfizer Investigational Site, Bucaramanga, Santander Department
  - Pfizer Investigational Site, Cali, Valle del Cauca Department
  - Pfizer Investigational Site, Calli, Valle del Cauca Department
- Pfizer Investigational Site, Monterrey, Nuevo León, Mexico
- Pfizer Investigational Site, Lima, Lima Province, Peru

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=VALA-0513-146&StudyName=A%20Multi-Center%2C%20Randomized%2C%20Double-Blind%2C%20Parallel%20Group%20Study%20To%20Compare%20The%20Efficacy%20And%20Tolerability%20Of%20Valdecoxib%20And%20Diclofena